CLINICAL TRIAL: NCT00765947
Title: A Twenty-four Week, Open-label, Non-comparative, Multi-center Study to Assess the Efficacy and Tolerability of an Aliskiren-based Treatment Algorithm in Patients With Mild to Moderate Hypertension.
Brief Title: Efficacy and Tolerability of an Aliskiren-based Treatment Algorithm in Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A2360
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Essential Hypertension ( Mild to Moderate)
Keywords: Essential Hypertension ( mild to moderate)
MeSH Terms: conditions — Essential Hypertension | interventions — aliskiren; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aliskiren-based regimen (Experimental): All pts starting on aliskiren 150 mg (uptitrated to aliskiren 300 mg), followed by the addition of HCTZ 12.5 mg (uptitrated to 25 mg) and amlodipine 5 mg (uptitrated to 10 mg), as necessary to achieve the Blood Pressure goal.
  Interventions: Drug: Aliskiren; Drug: Hydrochlorothiazide; Drug: Amlodipine

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 or 300 mg
Drug: Hydrochlorothiazide — Hydrochlorothiazide 12.5 or 25 mg
Drug: Amlodipine — Amlodipine 5 or 10 mg

SUMMARY:
This study will assess the efficacy of an aliskiren based treatment regimen in reaching blood pressure (BP) target in patients with mild to moderate hypertension. (defined as mean sitting Systolic Blood Pressure [msSBP] ≥ 140 mmHg and < 180 mmHg and/or mean sitting Diastolic Blood Pressure [msDBP] ≥ 90 and <110 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥ 18 years of age
* Patients with a diagnosis of mild to moderate hypertension at Visit 1
* All patients must have a msSBP ≥ 140 mmHg and < 180 mmHg and/or msDBP ≥ 90 mmHg and < 110 mmHg mmHg at Visit 3

Exclusion Criteria:

* Severe hypertension defined as msSBP ≥ 180 mmHg and/or msDBP ≥ 110 mmHg
* Secondary form of hypertension
* Current diagnosis of heart failure (NYHA Class II-IV)
* Current angina pectoris requiring pharmacological therapy (other than stable doses of oral or topical nitrates)
* Second or third degree heart block without a pacemaker
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia, atrial fibrillation or atrial flutter, during the 12 months prior to Visit 1

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Investigative Site, Paris, France
- Investigative Site, Budapest, Hungary
- Investigative Site, Bucharest, Romania
- Investigative Site, Bratislava, Slovakia

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren-based Regimen: Patients initiated treatment with aliskiren 150 mg (up-titrated to aliskiren 300 mg), followed by the addition of HCTZ 12.5 mg (up-titrated to 25 mg) and amlodipine 5 mg (up-titrated to 10 mg), as necessary to achieve the Blood Pressure goal.
Period: Overall Study
Arm/Group | Aliskiren-based Regimen
Started | 256
Completed | 232
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Aliskiren-based Regimen
Number analyzed (Participants) | 256
Age, Customized [Number; unit: participants]
  < 65 yrs | 203
  ≥ 65 yrs | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 143

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (Defined as Estimated Cumulative Control Rate) Reaching Blood Pressure Target in a Stepped Care, Aliskiren-based Regimen
Description: For non diabetic patients the Blood Pressure target is defined as mean sitting Systolic Blood Pressure [msSBP] < 140 mmHg and mean sitting Diastolic Blood Pressure [msDBP] < 90 mmHg and for diabetic patients the Blood Pressure target is mean sitting Systolic Blood Pressure [msSBP] < 130 mmHg and mean sitting Diastolic Blood Pressure [msDBP] < 80 mmHg.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren-based Regimen
Number analyzed (Participants) | 256
Percentage of participants | 86.12

2. Secondary Outcome: Percentage of Patients (Defined as Estimated Cumulative Control Rate) Reaching Blood Pressure Target in a Stepped-care, Aliskiren-based Regimen by Patient Subgroups of Mild and Moderate Hypertensive Patients, and Non-diabetic and Diabetic Patients.
Description: as for outcome 1
Time Frame: 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren-based Regimen
Number analyzed (Participants) | 256
Percentage of Participants
  Mild Hypertensive | 91.48
  Moderate Hypertensive | 79.24
  Non-diabetic | 92.74
  Diabetic | 72.58

3. Secondary Outcome: Changes From Baseline to Week 24 in Mean Sitting Systolic Blood Pressure [msSBP] and Mean Sitting Diastolic Blood Pressure [msDBP]
Time Frame: Baseline and Week 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren-based Regimen
Number analyzed (Participants) | 251
mm Hg
  msSBP | -25.33 (13.942)
  msDBP | -12.40 (9.371)

4. Secondary Outcome: Percent of Responders for Mean Sitting Systolic Blood Pressure [msSBP] and for Mean Sitting Diastolic Blood Pressure [msDBP]
Description: Response for mean sitting Systolic Blood Pressure [msSBP] is defined as a reduction of ≥ 20 mmHg from baseline or mean sitting Systolic Blood Pressure [msSBP] < 140 mmHg (non diabetics) or < 130 mmHg (diabetics). Response for mean sitting Diastolic Blood Pressure [msDBP] is defined as a reduction of ≥10 mmHg from baseline or mean sitting Diastolic Blood Pressure [msDBP] < 90 mmHg (non diabetic) or < 80 mmHg (diabetics).
Time Frame: 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren-based Regimen
Number analyzed (Participants) | 256
Percentage of Participants
  msSBP | 96.80
  msDBP | 97.78

ADVERSE EVENTS:
Groups:
- Aliskiren: Aliskiren treatment step
- Aliskiren + HCTZ: Aliskiren and HCTZ treatment step
- Aliskiren + HCTZ + Amlodipine: Aliskiren + HCTZ + Amlodipine treatment step
Arm/Group | Aliskiren | Aliskiren + HCTZ | Aliskiren + HCTZ + Amlodipine
Serious Adverse Events (participants affected / at risk) | 3/256 | 0/197 | 0/119
Other Adverse Events (participants affected / at risk) | 0/256 | 0/197 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=256) | Aliskiren + HCTZ (N=197) | Aliskiren + HCTZ + Amlodipine (N=119)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.